CLINICAL TRIAL: NCT05069545
Title: A Multi-centre Prospective Non-interventional Clinical Investigation Studying the Glycaemic Control in Patients With Type 1 Diabetes When Introducing a NovoPen® 6 for Treatment With Tresiba® (Insulin Degludec) & Fiasp® (Fast-acting Insulin Aspart) in a Real-world Setting
Brief Title: A Research Study Looking at How the Use of NovoPen® 6 for Treatment With Tresiba® & Fiasp® Affects the Blood Sugar Level in Patients With Type 1 Diabetes as Part of Local Clinical Practice
Acronym: CONNECT 1
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DV3325-4759; U1111-1255-5564 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tresiba + Fiasp using NovoPen 6 per local label: Participants will use Tresiba® and Fiasp® in NovoPen® 6 as prescribed to participants by the study doctor
  Interventions: Drug: Insulin degludec; Drug: Fast-acting insulin aspart

INTERVENTIONS:
Drug: Insulin degludec — Introducing a NovoPen® 6 to patients with type 1 diabetes mellitus (T1DM), who are already being treated with Tresiba® and Fiasp®
Drug: Fast-acting insulin aspart — Introducing a NovoPen® 6 to patients with type 1 diabetes mellitus (T1DM), who are already being treated with Tresiba® and Fiasp®

SUMMARY:
The purpose of this study is to collect information on how NovoPen® 6 works with Tresiba® & Fiasp® for treatment of people with type 1 diabetes and see if the use of NovoPen® 6 can help participants achieve better blood sugar levels.

Participants will use Tresiba® & Fiasp® in NovoPen® 6 as prescribed to participants by the study doctor.

NovoPen® 6 is a smart pen, which collects and stores the date and time of injections and number of units of insulin participants have taken.

NovoPen® 6 can transfer participants insulin dosing information to the mobile application, which participants use to see their continuous blood sugar level. This will allow participants to see their insulin doses along with continuous blood sugar level in the mobile application.

Participants will keep using their own continuous blood sugar monitoring device and the mobile application to see these data during the study.

The study will last for about 9-11 months. Participants will be asked to complete 2 questionnaires in this study. One questionnaire is about overall satisfaction of using a digital health solution and other is about quality of life. Participants will complete these questionnaires during their normally scheduled visit with the study doctor, on 2 separate occasions

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing consent.
* Diagnosed with T1DM (Type 1 Diabetes Mellitus) for above or equal to 1 year (365 days) at the time of signing consent.
* On treatment with Tresiba® for more than or equal to 1 month (30 days) and Fiasp® for for more than or equal to 3 months (90 days) at the time of signing consent.
* The decision to initiate the use of commercially available NovoPen® 6 as a part of treatment with Tresiba® and Fiasp® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Current user of a rtCGM (Real-Time Continuous Glucose Monitoring) or isCGM (Intermittent-scanning Continuous Glucose Monitoring) for greather than or equal to 2 months (60 days) of which the last 14 days must be on rtCGM or isCGM, which can integrate the data with diabetes treatment support solution from either Glooko or Abbott, at the time of signing consent.
* Willingness to continue using a rtCGM or isCGM for the duration of the study, which can integrate the data with diabetes treatment support solution from either Glooko or Abbott.
* Current user of a diabetes treatment support solution from either Glooko or Abbott, which can integrate the NovoPen® 6 injection data and the rtCGM/isCGM data, and willingness to continue using the same solution for the duration of the study.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given consent in this study.
* Treatment with any investigational drug within 30 days prior to enrolment into the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Use of any smart pen or smart cap for the diabetes treatment prior to the signing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will use Tresiba® and Fiasp® in NovoPen® 6 as prescribed to participants by the study doctor
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in time in range (3.9-10 mmol/L) | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM (Real-Time Continuous Glucose Monitoring) and isCGM data(Intermittent-scanning Continuous Glucose Monitoring))

SECONDARY OUTCOMES:
Change in time in hyperglycaemia/above range Level 1 (10.1 - 13.9 mmol/L) | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM and isCGM data)
Change in time in hyperglycaemia/above range Level 2 (greater than 13.9 mmol/L) | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM and isCGM data)
Change in time in hypoglycaemia/below range Level 1 (3.0-3.8 mmol/L) | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM and isCGM data)
Change in time in hypoglycaemia/below range Level 2 (below 3.0 mmol/L) | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM and isCGM data)
Change in mean glucose | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  mmol/L (Using available rtCGM and isCGM data)
Change in glucose variability (% coefficient of variability) | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM and isCGM data)
Change in Glucose Management Indicator | Baseline (Day -14 to Day 0) to End of Study (Day 280)
  Percentage change (absolute)
  (Using available rtCGM and isCGM data) (4The GMI is calculated from mean glucose as GMI (%) = 3.31 + 0.4306 [mean glucose mmol/L])
Change in HbA1c (Glycated haemoglobin) | Baseline (Week 0) to End of Study (Week 40)
  Percentage change (absolute) (Using HbA1c results based on blood tests)
T1-DDS (Diabetes Distress Scale for Adults with Type1 Diabetes), change in QoL (Quality of Life) | Baseline (Week 0) to End of Study (Week 40)
  Change (absolute) (Using T1-DDS questionnaire data)
DHSS (Digital Health Solution Satisfaction)-Patient | End of Study (Week 40)
  Total score (Using DHSS questionnaire for patient & HCP respectively)
DHSS-HCP(Health Care Professional) | End of Study (Week 40)
  Total score (Using DHSS questionnaire for patient & HCP respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (26):
- Belgium (6):
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - HUB - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc - Serv Endocrinologie - Diabétologie, Brussels
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Leuven - Endocrinology, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Denmark (4):
  - Aarhus Universitetshospital Diabetes og Hormonsygdomme, Aarhus N
  - Bispebjerg Hospital, IC-Forskning, Copenhagen
  - Medicinsk Afdeling B, Herning Centralsygehus, Herning
  - Regionshospitalet Silkeborg - Endokrinologisk afd., Silkeborg
- France (8):
  - Centre Hospitalier Universitaire de Caen Normandie- Cote de Nacre, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - hôpital Saint Joseph Saint Luc, Lyon
  - Centre Hospitalier Universitaire de Montpellier-Hopital Lapeyronie, Montpellier
  - Ap-Hp-Hopital Bichat-Claude Bernard-1, Paris
  - Hospices Civils de Lyon-Hopital Lyon Sud-2, Pierre-Bénite
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-2, Toulouse
  - Chru de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Sweden (8):
  - Diabetesmottagningen, Medicinkliniken, Södra Älvsborgs Sjukhus, Borås
  - Diabetesmottagningen, Södra Älvsborgs Sjukhus, Borås
  - Endokrinologiska kliniken, Malmö, Malmo
  - Medicinmottagning1 Universitetssjukhuset Örebro, Örebro
  - Centrum for Diabetes, Academical Specialist Centrum, Stockholm
  - Medicinkliniken Sundsv, Sundsvall
  - Uppsala universitetssjukhus, Uppsala
  - Frölunda Specialistsjukhus, Västra Frölunda

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com